CLINICAL TRIAL: NCT06358625
Title: Identification of Risk Factors for Brain Recurrence in Patients With HER2-positive Localised Breast Cancer
Acronym: CRANIUM
Status: Recruiting | Type: Observational
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-4-1-001
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: Metastases; Central Nervous System; Biopsy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER positive: The study will include an initial assessment and longitudinal and individual follow-up to identify the occurrence of clinical events of interest and to monitor the evolution of any tumour biomarkers on circulating tumour DNA.
  Interventions: Other: Pre-treatment biopsy

INTERVENTIONS:
Other: Pre-treatment biopsy — A breast biopsy is performed just before the "clip" is placed in the tumour and additional blood samples are performed.

SUMMARY:
HER2 gene amplification, detected in 20% to 30% of breast cancers, was a poor prognostic factor before the advent of anti-HER2 therapies. In the early 2000s, trastuzumab revolutionised the management of patients with HER2-positive (HER2+) breast cancer in the metastatic and localised stages of the disease.

At the time of diagnosis of metastatic disease, 7-11% of patients have brain metastases, with (70% of cases) or without symptoms (30% of cases). In the absence of brain metastases, 30% to 50% of patients will develop brain metastases within the first two years of treatment, depending on whether the disease is hormone receptor positive (HR+) or negative (HR-).

The presence of brain metastases is the most important prognostic factor. The neurological symptoms caused by the presence of these lesions, but also by the local treatments offered, affect patients' quality of life, although improvements in surgical and radiotherapy techniques have significantly reduced the need for particularly toxic whole brain radiotherapy.

International guidelines do not recommend systematic brain MRI in the absence of neurological symptoms, either in the adjuvant or metastatic stages of this disease. However, there may be a role for more systematic and earlier screening for cerebral recurrence, as single cerebral recurrences without extracranial involvement are common and the new anti-HER2 agents (i.e. tucatinib, an anti-HER2 tyrosine kinase inhibitor, and T-Dxd) have shown significant objective response rates in cerebral metastases.

To date, no clinical or histological prognostic factor (proliferation index, HR expression, etc.) has been used to identify a population of patients at high risk of cerebral relapse, allowing monitoring and treatment to be personalised.

New tools for these indications would significantly modify our clinical practice, allowing the identification of a subpopulation at high risk of cerebral recurrence, suitable for increased monitoring and therapeutic adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* be a female patient
* Patients with histologically proven HER2-positive invasive breast cancer (IHC 3+ or 2+ with positive SISH),
* Neoadjuvant chemotherapy and intra-tumour clips indicated at the multidisciplinary consultation meeting (RCP).
* Signed Informed Consent Form

Exclusion Criteria:

* pregnant or breast-feeding women
* Have had a haematoma requiring level II analgesics at the time of the diagnostic biopsy.
* Known coagulation disorders
* Individual deprived of liberty or placed under the authority of a tutor, or a currator
* Not be affiliated to a social security regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with HER2+ non-metastatic breast cancer treated at the CRLCC Eugène marquis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2031-06-06 (Estimated); Study Completion 2031-06-06 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic profile change of HER2+ primary breast tumours before any treatment | At inclusion
  comparison of the transcriptomic profile of HER2+ primary breast tumours before any treatment of patients who will develop brain metastases within 5 years with patients who will not develop them

SECONDARY OUTCOMES:
Transcriptomic profile change on circulating tumour DNA (ctDNA) | At baseline, Year 1; Year2; Year3, Year4; Year 5, at relapse
  High-throughput sequencing (NGS) of a panel of genes previously identified by transcriptomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LE DU, Dr, Principal Investigator — Centre de lutte contre le cancer Eugène Marquis
Locations (1):
- Centre de lutte contre le cancer Eugène Marquis, Rennes, France